CLINICAL TRIAL: NCT05578872
Title: A Phase 1/2 Study of ANV419 as Monotherapy or in Combination With Anti-PD-1 or Anti-CTLA-4 Antibody Following Anti-PD-1/Anti-PD-L1 Antibody Treatment in Patients With Unresectable or Metastatic Cutaneous Melanoma (OMNIA-1)
Brief Title: A Study of ANV419 Alone or in Combination With Approved Treatment in Patients With Cutaneous Melanoma (OMNIA-1).
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anaveon AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANV419-101
Record Dates: First submitted 2022-10-11; First posted 2022-10-13 (Actual); Results first posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Melanoma (Skin); Cutaneous Melanoma; Adult Disease; Advanced Solid Tumor; Metastatic Melanoma
Keywords: IL-2; ANV419; Cancer; Melanoma; OMNIA; Cutaneous; Metastatic; Anti-PD1
MeSH Terms: conditions — Melanoma; Disease; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ANV419 single agent, low dose (Experimental)
  Interventions: Drug: ANV419
- ANV419 single agent, high dose (Experimental)
  Interventions: Drug: ANV419

INTERVENTIONS:
Drug: ANV419 — ANV419 administered by intravenous (IV) infusion

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ANV419 monotherapy or the combination of ANV419 with anti-PD1 antibody or with anti-CTLA4 antibody in adult participants with advanced (unresectable or metastatic) cutaneous melanoma. The study has 3 parts. Part 1 to evaluate ANV419 in monotherapy and Parts 2 and 3 to evaluate ANV419 in combination with anti-PD1 antibody or anti-CTLA4 antibody. Parts 2 and 3 were not initiated, as the prespecified efficacy criteria to graduate to Part 2 were not met at the interim analysis of Part 1.

DETAILED DESCRIPTION:
The purpose of this multi-site, open-label, randomized, parallel arm, Phase 1/2 adaptive study is to evaluate the efficacy and safety of ANV419 as a monotherapy and in combination with anti-PD1 antibody or anti-CTLA4 antibody in patients aged 18 years or older with advanced Cutaneous Melanoma who have previously been treated with an anti-PD-1/anti-PD-L1 antibody.

ELIGIBILITY:
Inclusion Criteria:

* Must provide written informed consent for the study;
* Must be able to comply with the Protocol as judged by the Investigator;
* Are ≥18 years of age on day of signing informed consent;
* Have histologically confirmed Stage 3 (unresectable) or Stage 4 (metastatic) CM, as per the American Joint Committee on Cancer staging system, eighth edition;
* Have documented radiological progression on prior systemic therapy;
* Have previously received anti-PD-1/L1 as monotherapy or in combination. A maximum of 2 prior lines of systemic therapy is allowed for BRAF wild-type disease and a maximum of 3 prior lines of systemic therapy is allowed for BRAFV600 positive disease;
* Have measurable disease based on RECIST;
* Have a performance status of 0 or 1 on the ECOG Performance Status;
* Have adequate organ functions as defined per protocol;
* Female patients of childbearing potential must have a negative serum pregnancy test at the Screening Visit and a negative (urine or serum) pregnancy test within 72 hours prior to study Day 1. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required and must be negative for the patient to be eligible;
* Female patients who are not postmenopausal, and who have not undergone surgical sterilization, must agree to use highly effective methods of contraception during the treatment period and for 6 months after the last dose of study drug. They must also agree not to donate eggs (ova, oocytes) during the same timeframe; and
* Male patients with partners of childbearing potential must agree to use highly effective methods of contraception and barrier contraception (condom) during the treatment period and for 6 months after the last dose of study drug. They must also agree not to donate sperm during the same timeframe.

Exclusion Criteria:

* Have received investigational agent (including investigational device) within 4 weeks or an interval of 5 half-lives of the respective investigational agent prior to study Day 1, whichever is longer, with the exclusion of an anti-PD-1/anti-PD-L1 antibody given as either a single agent or non-CTLA-4 antibody containing combination (eg, anti-lymphocyte-activation gene 3 antibody);
* Have a known hypersensitivity to ANV419 or to any of the excipients, such as sucrose, histidine or polysorbate 80. For combination arms only: Have hypersensitivity to pembrolizumab or ipilimumab or any of their excipients;
* For combination arms only: Have previously discontinued ipilimumab, pembrolizumab or any other PD-1/PD-L1 inhibitors due to unacceptable drug-related toxicity (defined as toxicities that required second line immunosuppression, ie, not controlled by steroids alone);
* Have an LDH level of ≥2 × upper limit of normal;
* Have not recovered (ie, ≤Grade 1 or at baseline with the exception of alopecia or fatigue [up to Grade 2 allowed]) from AEs resulting from prior immunotherapies. Patients who have autoimmune AEs controlled by replacement therapy (ie, hypothyroidism) due to previous treatment are eligible provided replacement therapy has been initiated and toxicity has returned to Grade 1;
* Have not recovered (ie, ≤Grade 1 or at baseline) from toxicities due to a previously administered prior chemotherapy, targeted small molecule therapy, or radiation therapy; Note: If the patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study drug. Major surgery is defined as any surgery requiring entrance into a body cavity (eg, chest, abdomen, or brain), organ removal, normal anatomy alteration, or joint replacement. Minor surgery is defined as any surgery in which skin, mucosa, or connective tissue sections are altered (eg, biopsy, cataract, endoscopic procedures, etc).
* Have been diagnosed with uveal/ocular or mucosal melanoma;
* Have a known additional malignancy (including all in-situ carcinoma) that is progressing or required active treatment within ≤2 years prior to enrollment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that have undergone potentially curative therapy or in situ cervical cancer or patients who completed cancer-directed therapy and have no evidence of disease;
* Have active central nervous system metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to study Day 1 and any neurologic symptoms have returned to baseline or have been stable for at least 7 days), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study drug. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability;
* Have a diagnosis of immunodeficiency or is receiving immunosuppressive therapy within 7 days prior to study Day 1;
* Are receiving systemic steroid >10 mg of prednisone daily or equivalent or any other immunosuppressive medication at any dose level. Local steroid therapies (eg, otic, ophthalmic, intra-articular, or inhaled medications) are acceptable;
* Have an active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc) is not considered a form of systemic treatment;
* Have evidence of active, non-infectious pneumonitis;
* Have active (measurable) and uncontrolled (unresponsive to current therapy) infectious disease (bacterial, fungal, viral, or protozoic);
* Have a history of an acute coronary event (eg, myocardial infarction) within 3 months prior to study Day 1, uncontrolled and symptomatic coronary artery disease or congestive heart failure New York Heart Association Class III/IV;
* Have an average QTcF interval >470 msec at Screening;
* Have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or it is not in the best interest of the patient to participate, in the opinion of the treating Investigator;
* Have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study;
* Are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the Screening Visit through 6 months after the last dose of study drug;
* Are known to be human immunodeficiency virus (HIV) positive (or tests positive for HIV 1 or 2 at Screening), unless the following criteria are met: CD4+ lymphocyte count >350 µL; Had no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections within the past 12 months; Have been on established anti-retroviral therapy for at least 4 weeks; and Have an HIV viral load of <400 copies/mL prior to study Day 1. Note: Patients on strong cytochrome P450 (CYP)3A4 inhibitors or strong CYP3A4 inducers must be switched to an alternate effective anti-retroviral therapy regimen prior to study treatment or are excluded if regimen prior to study Day 1 cannot be altered.
* Have uncontrolled hepatitis B infection or hepatitis C infection; or Note: Patients with hepatitis B (positive hepatitis B surface antigen) who have controlled infection (serum hepatitis B virus DNA by polymerase chain reaction that is below the limit of detection and receiving anti-viral therapy for hepatitis B) are permitted. Patients with controlled infections must undergo periodic monitoring of hepatitis B virus DNA. Note: Patients with hepatitis C (positive hepatitis C virus antibody) who have controlled infection (undetectable hepatitis C virus RNA by polymerase chain reaction either spontaneously or in response to a successful prior course of anti-hepatitis C virus therapy) are permitted.
* Have received a live vaccine within 30 days of study Day 1; Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (eg, Flu-Mist®) are live attenuated vaccines, and are not allowed.
* For combination arms only: Have received solid organ or hematopoietic stem cell transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-12-16 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Gasal, MD, Study Director — Anaveon AG
Locations (25):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California San Diego, La Jolla, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Denver, Colorado
  - Northwestern University, Chicago, Illinois
  - HealthPartners Institute, Bloomington, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Atlantic Health System, Morristown, New Jersey
  - Virginia Cancer Specialists, Fairfax, Virginia
- France (6):
  - Centre Georges François Leclerc, Dijon
  - Centre Hospitalier Universitaire de Lille, Lille
  - CHU de Nantes, Nantes
  - AP-HP Hopital Saint-Louis, Paris
  - Gustave Roussy, Paris
  - CHU de Poitiers, Poitiers
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsmedizin der Johannes Gutenberg, Universität Mainz, Mainz
- Italy (3):
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori", Meldola
  - Istituto Nazionale Tumori IRCCS Fondazione G. Pascale, Napoli
  - Azienda Ospedaliero Universitaria Senese, Siena
- Spain (5):
  - Hospital Clinic de Barcelona, Barcelona
  - Centro Oncológico MD Anderson International España, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Universitary Hospital Virgen Macarena, Seville

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In line with the protocol, Parts 2 and 3 of the study were not initiated, as the prespecified efficacy criteria to graduate to Part 2 were not met during Part 1.
  No participants were enrolled in Parts 2 and 3 prior to the close of the study.
Period: Overall Study
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose
Started | 14 | 15
Completed | 0 | 0
Not Completed | 14 | 15
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Physician Decision | 1 | 2
Not completed — Progressive disease | 10 | 9
Not completed — Sponsor decision | 0 | 1
Not completed — Toxicity and Patient's decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose | Total
Number analyzed (Participants) | 14 | 15 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (14.15) | 59.8 (13.92) | 59.8 (13.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 8 | 16
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Monotherapy Dose Expansion: Objective Response Rate (ORR) as Defined by RECIST v1.1
Description: Proportion of participants with a complete response (CR) or partial response (PR) to treatment as defined by RECIST v1.1 (ORR = CR + PR)
Time Frame: Day 1 up to 12 months
Population: The efficacy population included patients who receive at least 1 dose of study drug and have at least 1 post-baseline tumor assessment. No patients achieved CR or PR.
Measure: Count of Participants; unit: Participants
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose
Number analyzed (Participants) | 14 | 14
Participants | 0 | 0

2. Secondary Outcome: Monotherapy Dose Expansion: Duration of Response (DOR) According to RECIST v1.1
Description: Time from first time measurement criteria are met for complete response (CR) or (PR) until the progressive disease or death.
Time Frame: Day 1 up to 12 months
Population: The efficacy population included patients who receive at least 1 dose of study drug and have at least 1 post-baseline tumor assessment. No patients achieved CR or PR so this outcome could not be assessed.
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Monotherapy Dose Expansion: Disease Control Rate (DCR) According to RECIST v1.1
Description: Percentage of participants who have achieved Complete Response (CR), Partial Response (PR) and Stable Disease (SD).
Time Frame: Day 1 up to 12 months
Population: The efficacy population included patients who receive at least 1 dose of study drug and have at least 1 post-baseline tumor assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose
Number analyzed (Participants) | 14 | 14
Participants | 5 | 7

4. Secondary Outcome: Monotherapy Dose Expansion: Progression-free Survival (PFS) According to RECIST v1.1
Description: Length of time participants lived with the disease without progressing (PD)
Time Frame: Day 1 up to 12 months
Population: The safety population is defined as all patients who receive at least 1 dose (or partial dose) of study drug(s).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose
Number analyzed (Participants) | 14 | 15
months | 2.2 [1.8 to 2.6] | 2.4 [1.4 to 4.4]

5. Secondary Outcome: Monotherapy Dose Expansion: Overall Survival (OS) Rate
Description: Proportion of participants who are alive at 6 months. This is an estimation based on Kaplan-Meier method.
Time Frame: Day 1 up to 6 months
Population: The Safety Population is defined as all patients who receive at least 1 dose (or partial dose) of study drug(s).
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose
Number analyzed (Participants) | 14 | 15
Proportion of participants | 0.8 [0.5 to 0.9] | 0.8 [0.5 to 0.9]

6. Secondary Outcome: Monotherapy Dose Expansion: Frequency of Treatment-Emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs.
Time Frame: Day 1 through study completion, an average of 3.7 months and a maximum of 14 months.
Population: The Safety Population is defined as all patients who receive at least 1 dose (or partial dose) of study drug(s)
Measure: Count of Participants; unit: Participants
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose
Number analyzed (Participants) | 14 | 15
Participants | 14 | 15

7. Secondary Outcome: Monotherapy Dose Expansion: Severity of TEAEs
Description: Number of participants with TEAEs Grade 3 or more.
Time Frame: Day 1 through study completion, an average of 3.7 months and a maximum of 14 months.
Population: The Safety Population is defined as all patients who receive at least 1 dose (or partial dose) of study drug(s)
Measure: Count of Participants; unit: Participants
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose
Number analyzed (Participants) | 14 | 15
Participants | 12 | 13

8. Secondary Outcome: Monotherapy Dose Expansion: Prevalence of Specific Anti-ANV419 Antibodies (ADA) in Blood
Description: Number of patients with positive ADA at baseline and end of study.
Time Frame: Day 1 through study completion, an average of 3.7 months
Population: The Immunogenicity Population is defined as all patients who receive at least 1 dose of study drug and have at least 1 evaluable immunogenicity sample.
Measure: Count of Participants; unit: Participants
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose
Number analyzed (Participants) | 14 | 15
Participants
  Prevalence of ADA positive at Baseline | 5 | 5
  Prevalence of ADA positive at End of Study | 12 | 5

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected during the full study period from the signing of the ICF through study completion, an average of 3.7 months and a maximum of 14 months.
Arm/Group | ANV419 Single Agent, Low Dose | ANV419 Single Agent, High Dose
All-Cause Mortality (participants affected / at risk) | 5/14 | 5/15
Serious Adverse Events (participants affected / at risk) | 10/14 | 11/15
Other Adverse Events (participants affected / at risk) | 14/14 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANV419 Single Agent, Low Dose (N=14) | ANV419 Single Agent, High Dose (N=15)
Thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Fistula of small intestine (Gastrointestinal disorders) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (5) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 6 (8) | 3 (5)
Spinal cord infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ANV419 Single Agent, Low Dose (N=14) | ANV419 Single Agent, High Dose (N=15)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 7 (17)
Coagulopathy (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (10)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 6 (16)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 2 (4)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 3 (4)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (8)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (3)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (9) | 9 (20)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Post-tussive vomiting (Gastrointestinal disorders) | 1 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (3) | 5 (23)
Asthenia (General disorders) | 8 (10) | 8 (12)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 3 (6) | 3 (15)
Face oedema (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (4) | 1 (1)
General physical health deterioration (General disorders) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 4 (4) | 2 (2)
Pain (General disorders) | 2 (3) | 0 (0)
Pyrexia (General disorders) | 5 (13) | 8 (21)
Swelling face (General disorders) | 0 (0) | 1 (2)
Cholestasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (2) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 7 (16) | 8 (20)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (4)
Urinary tract infection bacterial (Infections and infestations) | 1 (2) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (2) | 2 (3)
Alanine aminotransferase increased (Investigations) | 4 (11) | 8 (18)
Amylase increased (Investigations) | 2 (3) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (8) | 8 (19)
Bilirubin conjugated increased (Investigations) | 1 (1) | 1 (1)
Blood alkaline phosphatase decreased (Investigations) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 4 (4) | 3 (4)
Blood bilirubin increased (Investigations) | 3 (4) | 4 (7)
Blood calcium decreased (Investigations) | 0 (0) | 1 (1)
Blood chloride decreased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 5 (5)
Blood fibrinogen decreased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 2 (2) | 3 (3)
Blood phosphorus decreased (Investigations) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (3)
Blood urea increased (Investigations) | 0 (0) | 1 (2)
Blood uric acid increased (Investigations) | 1 (1) | 1 (1)
C-reactive protein increased (Investigations) | 2 (4) | 6 (8)
Fibrin D dimer increased (Investigations) | 1 (1) | 5 (8)
Gamma-glutamyltransferase increased (Investigations) | 4 (6) | 5 (17)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 2 (4) | 2 (7)
Lymphocyte count decreased (Investigations) | 1 (1) | 1 (2)
Lymphocyte count increased (Investigations) | 0 (0) | 3 (4)
Neutrophil count increased (Investigations) | 0 (0) | 1 (2)
Platelet count decreased (Investigations) | 1 (1) | 2 (2)
Platelet count increased (Investigations) | 0 (0) | 1 (1)
Protein total decreased (Investigations) | 0 (0) | 1 (5)
Protein urine present (Investigations) | 0 (0) | 1 (4)
Prothrombin level decreased (Investigations) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (4) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 1 (1) | 0 (0)
Urine protein/creatinine ratio increased (Investigations) | 0 (0) | 1 (4)
Weight decreased (Investigations) | 3 (4) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (3) | 3 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperchloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperferritinaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Hypophagia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (3)
Headache (Nervous system disorders) | 2 (4) | 2 (5)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 2 (3) | 2 (2)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 1 (2)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Granuloma skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (5)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3)
Vitiligo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must obtain Sponsor's written approval before any disclosure. Sponsor may delete confidential info, require edits, and delay release: 60-day review plus one-time patent embargo ≤ 90 additional days (total ≤ 150). Publication otherwise allowed after multicenter paper or 12 months post-study.

DOCUMENTS (2):
  • Study Protocol (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT05578872/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT05578872/SAP_001.pdf